CLINICAL TRIAL: NCT02397486
Title: The Impact of Pentoxifylline and Vitamin E on The Incidence and Severity of Radiotherapy- Induced Oral Mucositis and Dysphagia in Patients With Head and Neck Cancer
Brief Title: The Impact of Pentoxifylline and Vitamin E on Radiotherapy-induced Toxicity in Head & Neck Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rana Sayed Fouad, Assistant Lecturer- Clinical Pharmacy Department, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Ph.D 20
Record Dates: First submitted 2015-03-16; First posted 2015-03-25 (Estimated); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Pentoxifylline; Vitamin E; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): Platinum based concurrent chemoradiotherapy [cisplatin (100mg/m2) on day 1, 22 and 43 of Radiotherapy (at 2 Gy/ fraction to a dose of 70 Gy over 7 weeks] .
  Pentoxifylline 400 mg oral tablets twice daily for 7 weeks. Vitamin E 1000 mg oral capsules once daily for 7 weeks.
  Interventions: Drug: Pentoxifylline; Drug: Vitamin E; Drug: Cisplatin; Radiation: Radiation therapy
- Control Group (Active Comparator): Platinum based concurrent chemoradiotherapy [cisplatin (100mg/m2) on day 1, 22 and 43 of Radiotherapy (at 2 Gy/ fraction to a dose of 70 Gy over 7 weeks] .
  Interventions: Drug: Cisplatin; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Pentoxifylline
  Other Names: Trental
  Arms: Intervention Group
Drug: Vitamin E
  Arms: Intervention Group
Drug: Cisplatin
Radiation: Radiation therapy

SUMMARY:
The purpose of this study is to determine whether pentoxifylline and vitamin E are effective in prevention of radiotherapy- induced toxicity in head and neck cancer patients treated with concurrent chemoradiotherapy.

DETAILED DESCRIPTION:
This is a randomized controlled prospective study of pentoxifylline and vitamin E given on daily basis throughout the period of concurrent chemoradiotherapy to patients with carcinoma of the head and neck. All patients will be followed up to 90 days since the first day of treatment. The incidence and severity of adverse events will be assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Measurable disease
* Patients with squamous cell carcinoma of the head and neck eligible for treatment with concurrent chemo- radiotherapy
* Able to understand and willing to sign a written informed consent document

Exclusion Criteria:

* Pregnant or lactating women, since imaging cannot be done in this setting.
* Patients treated with vitamin E and/ or pentoxifylline for any other indication
* Patients with recent cerebral and/or retinal hemorrhage
* Patients who have previously exhibited intolerance to pentoxifylline or methylxanthines such as caffeine, theophylline, and theobromine.
* Patients treated with oral anticoagulants.
* Absolute neutrophil count ≤1.5×109/L
* Platelets ≤100×109/L
* AST ≥ 2.5 X institutional upper limit normal (ULN)
* Serum creatinine ≥ 1.5 mg% for males & 1.4 mg% for females
* Serum bilirubin ≥ 1.5X institutional upper limit normal (ULN)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-05-02 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of radiotherapy-induced toxicity | 90 days since start of treatment
  weekly follow-up for recording radiotherapy-induced toxicity occurrence.weekly reported toxicities will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03

SECONDARY OUTCOMES:
Duration of grade 3 or 4 radiotherapy-induced toxicity | 90 days since start of treatment
Patients' response to concurrent chemo-radiotherapy (objective response rate) | 63 days since start of treatment
  the effect of pentoxifylline and vitamin E on the
incidence and grade of pentoxifylline and vitamin E- related adverse events (National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03) | 90 days since start of treatment
  Adverse events induced by intervention drugs will be assessed according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03
Number of patients with unplanned breaks in radiotherapy | 49 days since start of treatment
Total dose of opioid analgesics required | 90 days since start of treatment
Functional oral intake score | 90 days since start of treatment
Patients' quality of life assessed using the validated Arabic version of the EuroQol-5D-3L questionnaire | 90 days since start of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sayed R, El Wakeel L, Saad AS, Kelany M, El-Hamamsy M. Pentoxifylline and vitamin E reduce the severity of radiotherapy-induced oral mucositis and dysphagia in head and neck cancer patients: a randomized, controlled study. Med Oncol. 2019 Nov 21;37(1):8. doi: 10.1007/s12032-019-1334-5. PMID 31748905